CLINICAL TRIAL: NCT03661502
Title: Effect of Variable Volume Ventilation on Lung Compliance During Mechanical Ventilation.
Brief Title: Effect of Variable Volume Ventilation on Lung Compliance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Jan Mulier, head of dep anesthesia & intensive care, AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JPM 2018 VVV
Record Dates: First submitted 2018-09-04; First posted 2018-09-07 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Lung Injury
MeSH Terms: conditions — Lung Injury

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- variable tidal volume ventilation (VVV) (Experimental): the intervention is using a ventilation mode with variable tidal volume. The average tidal volume is 6 ml/kg and respiratory rate adapted to reach an end tidalCO2 concentration between 30 and 50 mmHg. Lung recruitment is given when dynamic lung compliance drops below 40. No drug is given. No other treatment or intervention is given.
  Interventions: Device: VVV
- Pressure controlled ventilation (PCV) (Experimental): the intervention is using ventilation mode with constant pressure and constant tidal volume. The tidal volume is 6 ml/kg and respiratory rate is adapted to reach end tidal CO2 concentrations between 30 and 50 mmHg. Lung recruitment is given when dynamic lung compliance drops below 40. No drug is given. No other treatment or intervention is given.
  Interventions: Device: PCV

INTERVENTIONS:
Device: VVV — ventilation mode with variable tidal volume is chosen. the average tidal volume is 6 ml/kg and respiratory rate adapted to reach end tidal con between 30 and 50 mmHg
  Arms: variable tidal volume ventilation (VVV)
Device: PCV — ventilation mode with constant tidal volume is chosen. the tidal volume is 6 ml/kg and respiratory rate adapted to reach end tidal con between 30 and 50 mmHg
  Arms: Pressure controlled ventilation (PCV)

SUMMARY:
Randomized controlled trial comparing low inspiratory and expiratory flow during variable volume ventilation with a constant volume decelerating flow (pressure controlled volume guarantee) ventilation.

DETAILED DESCRIPTION:
Randomized controlled trial comparing low inspiratory and expiratory flow during variable volume ventilation (VVV) with a constant volume decelerating flow (PCV pressure controlled volume guarantee) ventilation.

After anesthesia induction patients are VVV or PCV ventilated with a positive end expiratory pressure (PEEP) of 10 cm H2O. Average tidal volume is set at 6 ml/kg and end tidal CO2 is kept between 30 and 50 mmHg in both groups by adapting breaths per minute between 10 and 16. I/E ratio is set at 1/1 in VVV and at the standard ½ in PCV.

Dynamic lung compliance is measured before and during pneumoperitoneum. If dynamic lung compliance is less than 40 or decreases below 40 a first lung recruitment (10 sec of 30 up to 40 cmH2O) is given till dyn compliance rises above 40.

Dynamic lung compliance is further monitored and when value decreases again below 40, a new lung recruitment (LRM) is given and the PEEP is increased to 15 cm H2O after the second LRM.

All patients get an opioid free general anesthesia with anti inflammatory agents and deep NMB with full reversal at end of surgery.

The moment and number of LRM performed after induction of anesthesia with the averaged reached lung compliance is used to compare both ventilation methods.

The oxygen saturation without oxygen at arrival of PACU and the need for oxygen when saturation drops below 95 % are compared between both groups.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic bariatric surgery requiring mechanical ventilation

Exclusion Criteria:

* lung disease requiring oxygen before anesthesia
* emergence procedure
* spontaneous or assisted ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of lung recruitments required to keep dynamic lung compliance above 40. | during mechanical ventilation under general anesthesia between 1 and 3 hours. No outcome measurements are measured after 3 hours.
  Measuring dynamic lung compliance during mechanical ventilation. When it drops below 40 a lung recruitment is done with increase of PEEP to maximum 15 cmH2O.

SECONDARY OUTCOMES:
Oxygen saturation at arrival of PACU without oxygen therapy. | during stay in PACU being between 1 and 4 hours post operative of the same day. No outcome measurements are measured after 4 hours.
  oxygen saturation on arrival of PACU without giving oxygen I measured and compared between both groups

CONTACTS AND LOCATIONS:
Overall Officials: Marc Lanckneus, Study Chair — AZ Sint-Jan AV
Locations (1):
- Azsintjan, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No